CLINICAL TRIAL: NCT03564418
Title: Ultrasound-Guided Thermocoagulation of Medial Nerve Branch in Lumbar Facet Joints Pain. Effectiveness and Benefits of a Non Irradiating Technique.
Brief Title: Ultrasound-Guided Thermocoagulation of Medial Nerve Branch in Lumbar Facet Joints Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2017/552
Record Dates: First submitted 2018-06-11; First posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Low Back Pain; Facet Joint Pain; Facet Syndrome of Lumbar Spine; Chronic Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Prospective, Controlled, Open trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-Guided Thermocoagulation of Lumbar facet joints (Active Comparator): Prone position: Thanks to a high-resolution ultrasound and a 5 MHz curved probe, we will use the ultrasound technique described by Greher et al to reach the target points. Then, in order to check the correct positioning of the needles, we will inject 1 ml of a solution of contrast medium (omnipaque® 300 mg / ml of Iohexol) to observe them using the standard Fluoroscopic method. Wrongly positioned needles will be correctly repositioned and these patients will be excluded from ODI and VAS scale statistics.
  Interventions: Procedure: Ultrasound-Guided Thermocoagulation of Lumbar facet joints
- Fluoroscopy-Guided Thermocoagulation of Lumbar facet joints (Active Comparator): Prone position: We will use the standard fluoroscopic method to reach the target points. (maximum three levels, same side). Then, in order to check the correct positioning of the needles, we will inject 1 ml of a solution of contrast medium (omnipaque® 300 mg / ml of Iohexol). The correct location being the superolateral edge of the lateral facet and the diffusion of the contrast material at the level of the medial branch observed thanks to an anteroposterior radioscopic view. Then the location of the needles is confirmed by a lateral radioscopic view.
  Interventions: Procedure: Fluoroscopy-Guided Thermocoagulation of Lumbar facet joints

INTERVENTIONS:
Procedure: Ultrasound-Guided Thermocoagulation of Lumbar facet joints — Prone position: Thanks to a high-resolution ultrasound and a 5 MHz curved probe, we will use the ultrasound technique described by Greher et al to reach the target points.
  Then, in order to check the correct positioning of the needles, we will inject 1 ml of a solution of contrast medium (omnipaque® 300 mg / ml of Iohexol) to observe them using the standard Fluoroscopic method. Wrongly positioned needles will be correctly repositioned and these patients will be excluded from ODI and VAS scale statistics.
  To ensure the effectiveness of the injury by thermocoagulation, sensory electrical stimulation is performed to confirm that the needle is close to the posterior ramus (50Hz, 0-3 volts) and another electrical stimulation is performed to confirm that there is no motor stimulation (2Hz, 0-3 volts). After injecting 1 ml of 2% linisol® through the needle, denervation of the facet will be performed with an electrode at 68 ° C for 90 seconds.
  Arms: Ultrasound-Guided Thermocoagulation of Lumbar facet joints
Procedure: Fluoroscopy-Guided Thermocoagulation of Lumbar facet joints — Prone position: We will use the standard fluoroscopic method to reach the target points. (maximum three levels, same side). Then, in order to check the correct positioning of the needles, we will inject 1 ml of a solution of contrast medium (omnipaque® 300 mg / ml of Iohexol). The correct location being the superolateral edge of the lateral facet and the diffusion of the contrast material at the level of the medial branch observed thanks to an anteroposterior radioscopic view. Then the location of the needles is confirmed by a lateral radioscopic view.
  To ensure the effectiveness of the injury by thermocoagulation, sensory electrical stimulation is performed to confirm that it is close to the posterior ramus (50Hz, 0-3 volts) and another electrical stimulation is performed to confirm that there is no motor stimulation (2Hz, 0-3 volts). After injecting 1 ml of 2% linisol® through the needle, denervation of the facet will be performed with an electrode at 68 ° C for 90 seconds.
  Arms: Fluoroscopy-Guided Thermocoagulation of Lumbar facet joints

SUMMARY:
We propose here to evaluate the precision of lumbar thermocoagulation performed under a transverse ultrasound approach by performing a fluoroscopic control once the needle in the desired position. The effectiveness of the technique will be assessed by measuring different pain and disability scores at six weeks post-thermocoagulation: the Visual analogue pain Scale score (VAS) and the Oswestry disability score (ODI) will be collected, compared to that of the conventional fluoroscopic technique.

DETAILED DESCRIPTION:
Low back pain affects 70 to 80% of people at least once in their lives. They have considerable socio-economic repercussions and represent the leading medical cause of work stoppage, at around 25% .1

The articular pain between the lumbar vertebrae, called facet joints pain, represent between 15 and 45% of all low back pain and their manifestations are grouped under the name of facet syndrome including localized pains at the lumbar level as well as pains referred to the gluteal, trochanteric, inguinal and lateral and posterior region of the thigh. 2-5 The thermocoagulation of the roots innervating the lumbar facets consists in creating a lesion of the nerve roots innervating these articulations in order to block the transmission of the pain.

According to many studies this technique gives good results in 70 to 80% of the cases with an improvement around 71% to more than six months. 6 A recent Meta-analysis involving 454 patients also shows a significant improvement at 12 months of thermocoagulation versus placebo and even versus epidural lumbar. 7

To date, Lumbar Thermocoagulation are still mostly performed under fluoroscopic control by injection of contrast. This technique have proved this effectiveness, but have significant disadvantages, such as the irradiation of the patient as well as that of the practitioner because of the number of daily acts performed and its cost.

For its part, ultrasound is easily available, easy to use, represents a lower cost, and the lack of irradiation. The technique to reach the lumbar facet joints with sonography is pretty well described and known for many years. 8

We propose here to evaluate the precision of lumbar thermocoagulation performed under a transverse ultrasound approach by performing a fluoroscopic control once the needle in the desired position. The effectiveness of the technique will be assessed by measuring different pain and disability scores at six weeks post-thermocoagulation: the Visual analogue pain Scale score (VAS) and the Oswestry disability score (ODI) will be collected, compared to that of the conventional fluoroscopic technique.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18.
* Facet Syndrome.
* Symptomatology superior than 3 mounths.
* A failure of conservative treatement (drugs, physiotherapy...)
* Partial improvement after two lumbar facet infiltrations.

Exclusion Criteria:

* Allergy to any of the constituents of the infiltrated product, or to the contrast medium
* Unstable medical condition: cardiac, respiratory, endocrine (uncontrolled diabetes)
* Local infection (cutaneous, perimedullary / spinal) or systemic.
* Coagulopathy (platelets <50000 / mm3, Prothrombin time <60%, INTernational normalized ratio> 1.5), anticoagulant or antiplatelet therapy treatment other than aspirin.
* Lumbar arthrodesis.
* Neurological condition affecting motor function (Stroke, Parkinson...)
* Pregnant woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of needle placement under ultrasound guidance | Before infiltration
  Good position: G. Wrong position: W.

SECONDARY OUTCOMES:
Visual Analogue scale | Baseline, 6 weeks
  0/10 (minimum) to 10/10 (maximum)
Oswestry Disability index | Baseline, 6 weeks
  % out of 50 questions (0/50= 0% to 50/50= 100%)

CONTACTS AND LOCATIONS:
Overall Officials: Luc Van Obbergh, PhD, Study Director — Chief of staff Anesthesiology
Locations (1):
- sebastian Jorquera Vasquez, Brussels, Anderlecht, Belgium

REFERENCES:
- [Background] Rimmalapudi V, Buchalter J, Calodney A. Radiofrequency Denervation for Chronic Low Back Pain. JAMA. 2017 Dec 12;318(22):2255-2256. doi: 10.1001/jama.2017.16378. No abstract available. PMID 29234798
- [Background] Cohen SP, Raja SN. Pathogenesis, diagnosis, and treatment of lumbar zygapophysial (facet) joint pain. Anesthesiology. 2007 Mar;106(3):591-614. doi: 10.1097/00000542-200703000-00024. PMID 17325518
- [Background] Fukui S, Ohseto K, Shiotani M, Ohno K, Karasawa H, Naganuma Y. Distribution of referred pain from the lumbar zygapophyseal joints and dorsal rami. Clin J Pain. 1997 Dec;13(4):303-7. doi: 10.1097/00002508-199712000-00007. PMID 9430810
- [Background] Lee CH, Chung CK, Kim CH. The efficacy of conventional radiofrequency denervation in patients with chronic low back pain originating from the facet joints: a meta-analysis of randomized controlled trials. Spine J. 2017 Nov;17(11):1770-1780. doi: 10.1016/j.spinee.2017.05.006. Epub 2017 May 30. PMID 28576500
- [Result] Greher M, Scharbert G, Kamolz LP, Beck H, Gustorff B, Kirchmair L, Kapral S. Ultrasound-guided lumbar facet nerve block: a sonoanatomic study of a new methodologic approach. Anesthesiology. 2004 May;100(5):1242-8. doi: 10.1097/00000542-200405000-00028. PMID 15114223
- [Result] Jung H, Jeon S, Ahn S, Kim M, Choi Y. The validation of ultrasound-guided lumbar facet nerve blocks as confirmed by fluoroscopy. Asian Spine J. 2012 Sep;6(3):163-7. doi: 10.4184/asj.2012.6.3.163. Epub 2012 Aug 21. PMID 22977695
- [Result] Kim D, Choi D, Kim C, Kim J, Choi Y. Transverse process and needles of medial branch block to facet joint as landmarks for ultrasound-guided selective nerve root block. Clin Orthop Surg. 2013 Mar;5(1):44-8. doi: 10.4055/cios.2013.5.1.44. Epub 2013 Feb 20. PMID 23467334